CLINICAL TRIAL: NCT07310004
Title: Virtual Reality vs. Music Relaxation for Reducing Anxiety and Pain During Breast Biopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-6080
Record Dates: First submitted 2025-02-19; First posted 2025-12-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Biopsy; Anxiety; Pain
Keywords: Breast Biopsy; Virtual Reality; Mindfulness; Pain Reduction; Anxiety Reduction
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with three parallel groups: VR intervention, music relaxation, and standard care. Participants will be randomized in a 1:1:1 ratio, and interventions will last for the duration of the biopsy procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Intervention (Experimental): Patients will wear a Virtual Reality (VR) headset during the breast biopsy. They will use the CS VR Mindful Meditation App. Anxiety and pain will be measured using validated scales, and an optional physiological marker may be collected to assess stress levels. Participants will also be asked about their satisfaction with the intervention received, along with procedure-specific questions.
  Interventions: Other: Virtual Reality (VR) Mindful App
- Music Intervention (Active Comparator): Patients will listen to standard calming music during the breast biopsy from the computer/speakers in the room. Anxiety and pain will be measured using validated scales, and an optional physiological marker may be collected to assess stress levels. Participants will also be asked about their satisfaction with the intervention received, along with procedure-specific questions.
  Interventions: Other: Standard Calming Music
- No Intervention (No Intervention): Patients will have no intervention and complete the breast biopsy as standard of care. Anxiety and pain will be measured using validated scales, and an optional physiological marker may be collected to assess stress levels. Participants will also be asked about their satisfaction with the intervention received, along with procedure-specific questions.

INTERVENTIONS:
Other: Virtual Reality (VR) Mindful App — Patients will wear a Virtual Reality (VR) headset and use an application called CS VR Mindful Meditation App.
  Arms: VR Intervention
Other: Standard Calming Music — Patients will listen to standard calming music played in the room.
  Arms: Music Intervention

SUMMARY:
This study aims to compare the effectiveness of a Virtual Reality (VR) application computer simulation [(CS) VR Mindful Meditation App')] versus music relaxation in reducing anxiety and pain in women undergoing breast biopsies. Participants will be randomized into three groups: VR, music relaxation, or standard care. Anxiety and pain will be measured using validated scales, and an optional physiological marker may be collected to assess stress levels. Participants will also be asked about their satisfaction with the intervention received, along with procedure-specific questions.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older.
* Scheduled for an ultrasound-guided or stereotactic breast biopsy.
* Capable of understanding and providing informed consent.

Exclusion Criteria:

* Individuals with a history of epilepsy, motion sickness, or severe cognitive impairment (for the VR group).
* Use of anxiolytic medication immediately prior to the biopsy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety | perioperatively/periprocedurally
  Pre- and post-procedure anxiety will be measured using the State-Trait Anxiety Inventory (STAI). The scale uses a four point Likert scale ranging from "not at all" to "very much so." The score range is from 20-80 with a higher score indicating more anxiety. The change in anxiety scores (pre- to post-procedure) will be compared across the three groups (VR, music relaxation, and control).
Pain Level | perioperatively/periprocedurally
  Pain will be measured using the Visual Analog Scale (VAS) before and after the procedure. The scale is a subjective measure where individuals mark pain intensity on a 100mm line. typically from "no pain" (0) to "wort possible pain" (100). Higher score is worse. The change in pain scores (pre- to post-procedure) will be analyzed. The

SECONDARY OUTCOMES:
Physiological Markers | During Biopsy
  Heart Rate Variability (RR intervals) may be recorded during the biopsy as an objective marker of anxiety and stress. This will be an optional measure and will require the patient to wear either a Polar H10 Heart Rate Sensor below the breast or a Heart Rate Sensor on the arm during the procedure.
Satisfaction Scores | immediately after the intervention/procedure/surgery
  For participants in the VR and music relaxation groups, a 5-point Likert scale will measure their satisfaction with the intervention. The "Intervention Satisfaction Question" asks "How satisfied were you with the intervention you received?", with 1 being "Not at all satisfied" and 5 being "Extremely satisfied". In this scale, a higher score means a better outcome. There is also the option for "I received no intervention."

CONTACTS AND LOCATIONS:
Locations (1):
- Westwood, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided